CLINICAL TRIAL: NCT03408236
Title: Randomized, Double-blind, Active-controlled, Multicenter, Phase I/III Clinical Trial to Evaluate the Safety and Efficacy of Botulax® as Compared to Botox® in Subject With Moderate to Severe Crow's Feet Lines
Brief Title: Evaluate the Safety and Efficacy of Botulax® as Compared to Botox® in Subject With Moderate to Severe Crow's Feet Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HG-BOTCFL-III1
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Crow's Feet Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulax (Experimental): Single dose
  Interventions: Drug: Botulinum toxin type A
- Botox (Active Comparator): Single dose
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Experimental
  Other Names: Botulax
  Arms: Botulax
Drug: Botulinum toxin type A — Active Comparator
  Other Names: Botox
  Arms: Botox

SUMMARY:
To determine the efficacy and safety of Botulax® in treatment of crow's feet line

DETAILED DESCRIPTION:
1. Allocation: Randomized
2. Masking: Double Blind

ELIGIBILITY:
Inclusion Criteria:

* Male or female of at least 19 to 65 years old
* Bilaterally symmetrical moderator-to-severe CFL at maximum smile on the FWS as rated by the investigator

Exclusion Criteria:

* Subject with hypersensitivity to the investigational products or their components
* Female subject who are pregnant or lactating
* Subject who are unable to communicate or follow the instructions
* Subject who are not eligible for this study based on the judgment of an investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Facial Wrinkle Scale(FWS) severity of crow's feet lines(CFL) at maxium smile as assessed by investigators | 4weeks
  The Investigator assessed the severity of the patient's Crow's Feet lines at maximum smile using the 4-point Facial Wrinkle Scale where 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a score of none or mild at Day 30 is reported as assessed by investigators

CONTACTS AND LOCATIONS:
Locations (1):
- Hugel, Seoul, South Korea

REFERENCES:
- [Derived] Yoo KH, Park SJ, Han HS, Won CH, Lee YW, Kim BJ. Randomized, double-blind, active-controlled, multicentre, phase III clinical trial with two stages to assess the safety and efficacy of letibotulinum toxin a vs. onabotulinum toxin a for subjects with moderate to severe crow's feet. J Eur Acad Dermatol Venereol. 2021 Jul;35(7):1587-1594. doi: 10.1111/jdv.17217. Epub 2021 Apr 12. PMID 33721365